CLINICAL TRIAL: NCT01699529
Title: Multi-electrode Radiofrequency Renal Denervation System Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10058715DOC
Record Dates: First submitted 2012-09-21; First posted 2012-10-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Denervation (Experimental)
  Interventions: Device: Medtronic Multi-electrode Radiofrequency (RF) Renal Denervation system

INTERVENTIONS:
Device: Medtronic Multi-electrode Radiofrequency (RF) Renal Denervation system — The Medtronic Multi-electrode Radiofrequency Renal Denervation System is comprised of a single-use, disposable catheter and a reusable generator.

SUMMARY:
This is a prospective, single-arm, non-randomized and open label feasibility study. The study is intended to evaluate safety and efficacy of multi-electrode radiofrequency renal denervation in patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥ 18 and ≤ 80 years old.
* Individual has an office systolic blood pressure of 160 mmHG or greater (≥ 150 mmHg for Type 2 diabetics) based on an average of 3 office/clinic blood pressure readings
* Individual is adhering to a stable medication regimen including ≥ 3 anti-hypertensive medications(preferred that one is a diuretic) for a minimum of two weeks prior to screening.

Exclusion Criteria:

* Individual has an estimated glomerular filtration rate (eGFR) of < 45 mL/min/1.73 m2
* Individual has type 1 diabetes mellitus
* Individual requires chronic oxygen support or mechanical ventilation (e.g., tracheostomy, CPAP, BiPAP) other than nocturnal respiratory support for sleep apnea.
* Individual has primary pulmonary hypertension.
* Individual is pregnant, nursing or planning to be pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Acute safety as measured by procedural complications | 1 month

SECONDARY OUTCOMES:
Change in Office Systolic Blood Pressure | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Whitbourn, MD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (4):
- Australia (3):
  - Alfred Hospital, Melbourne, Victoria
  - St. Vincent's Hospital Melbourne, Melbourne, Victoria
  - Epworth Hospital, Melbourne, Victoria
- Wellington Hospital, Wellington, Wellington Region, New Zealand

REFERENCES:
- [Derived] Whitbourn R, Harding SA, Walton A. Symplicity multi-electrode radiofrequency renal denervation system feasibility study. EuroIntervention. 2015 May;11(1):104-9. doi: 10.4244/EIJV11I1A18. PMID 25982652